CLINICAL TRIAL: NCT06573073
Title: Evaluation of Clinical Performance and IVD Test of LifeOS Digital PCR Liquid Biopsy Kits for EGFR T790M Mutation
Status: Recruiting | Type: Observational
Sponsor: LifeOS Genomics Corporation (Industry)
Collaborators: National Taiwan University (Other); National Taiwan University Hospital (Other); Chung Shan Medical University (Other); Chang Gung Memorial Hospital (Other); Tri-Service General Hospital (Other); Far Eastern Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202405068DSA
Record Dates: First submitted 2024-08-11; First posted 2024-08-27 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-08

CONDITIONS: Non Small Cell Lung Cancer; EGFR T790M
Keywords: Liquid biopsy; digital Polymerase Chain Reaction (PCR); EGFR T790M
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Biospecimen Retention: Samples With DNA — plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- NSCLC with EGFR mutation

SUMMARY:
Liquid biopsy plays a pivotal role in cancer therapeutics, encompassing critical applications such as early cancer detection, disease progression monitoring, and tailored treatment plan formulation, heralded as a pivotal avenue for the future of cancer management. Established in 2015, LifeOS Genomics Co., Ltd. stands among the select few domestic enterprises pioneering the autonomous development of digital Polymerase Chain Reaction (PCR) technology. The company's automated nucleic acid amplification quantitative analysis platform (QLoci™ md1000 Analyzer) demonstrates outstanding proficiency, featuring sixty thousand wells per PCR chip. Integrating digital PCR technology, it elevates analytical sensitivity beyond 0.1%. LifeOS commissioned the Core Laboratory of Pharmacogenomics at the National Taiwan University to conduct clinical validation assessments for their developed "EGFR T790M Mutation Detection Assay Kit." This assay kit secured official registration by the Taiwan Food and Drug Administration (TFDA) as a Laboratory Developed Test (LDT) in 2023, permitting the issuance of medical testing reports.

This initiative aims to validate the detection capabilities of LifeOS Genomics Co., Ltd.'s "EGFR T790M Mutation Detection Assay Kit" prospectively clinically in clinical lung cancer patient plasma samples, addressing unmet clinical needs for early cancer detection, disease progression monitoring, and aiding physicians in diagnosis and pharmacotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. aged ≥18 years old.
2. Patients with Stage IIIB or IV non-small cell lung cancer (NSCLC) with EGFR mutations.

Exclusion Criteria:

1. Pregnant women.
2. Any condition that, in the opinion of the doctors, may pose a severe risk to the patient or interfere with trial results or participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Late stage NSCLC patients with EGFR activating mutations
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-09-06 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Concordance in detecting EGFR T790M using the LifeOS EGFR T790M cfDNA Detection Kit and the cobas® EGFR Mutation Test v2. | 5 years
  The primary endpoint is to assess the concordance between the LifeOS EGFR T790M cfDNA Detection Kit and the cobas® EGFR Mutation Test v2 in detecting the presence of EGFR T790M in cfDNA from plasma.

SECONDARY OUTCOMES:
Sensitivity of the LifeOS EGFR T790M cfDNA Detection Kit relative to the cobas® EGFR Mutation Test v2. | 5 years
  The secondary endpoint is to assess the sensitivity between the LifeOS EGFR T790M cfDNA Detection Kit and the cobas® EGFR Mutation Test v2 in detecting the presence of EGFR T790M in cfDNA from plasma.
Specificity of the LifeOS EGFR T790M cfDNA Detection Kit relative to the cobas® EGFR Mutation Test v2. | 5 years
  The secondary endpoint is to assess the specificity between the LifeOS EGFR T790M cfDNA Detection Kit and the cobas® EGFR Mutation Test v2 in detecting the presence of EGFR T790M in cfDNA from plasma.

CONTACTS AND LOCATIONS:
Overall Officials: Sung-Liang Yu, PhD, Principal Investigator — National Taiwan University
Locations (1):
- National Taiwan University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No